CLINICAL TRIAL: NCT06562465
Title: Research on Prevention and Intervention of Overweight and Obesity in Preschool Children
Brief Title: Prevention and Intervention of Overweight and Obesity in Preschool Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chen Li (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other); China Soong Ching Ling Foundation (Other)
Responsible Party: Sponsor-Investigator, Chen Li, Associate Professor, Director, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OABIPC
Record Dates: First submitted 2024-07-11; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Overweight and Obesity
Keywords: Diet management; sports management; overweight; obesity; preschool children
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Recruit at least 174 overweight and obese children from kindergartens with a population of 200 or more in Chongqing, and recruit them in the order of screening and informed consent until they are fully recruited. Divided into intervention group and blank control group based on kindergarten.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The overweight and obese children aged 3-6 years old,receive dietary and exercise management, combined reward support mechanisms.
  Interventions: Procedure: dietary and exercise management
- Control group (Active Comparator): The overweight and obese children aged 3-6 years old only receive basic health guidance,do not receive dietary and exercise management nor combined reward support mechanisms like experimental group.
  Interventions: Procedure: no dietary and exercise management

INTERVENTIONS:
Procedure: dietary and exercise management — Dietary and exercise management: dietary management by providing tailored recipes, health education lectures, science competitions, etc；exercise management:develop weekly and monthly exercise plans for children of different ages, and have physical education teachers lead them in exercising.
  Arms: Experimental group
Procedure: no dietary and exercise management — NO dietary and exercise management:do not implement dietary and exercise management related to the experimental group
  Arms: Control group

SUMMARY:
Obesity is an important public health problem, which is directly related to the risk of childhood complications and the increase of incidence rate and mortality of adult complications. The consequences are more serious than malnutrition such as low weight. Since the 1980s, the obesity rate among children in China has gradually increased. Currently, overweight and obesity are important health issues for children in rural and urban areas of China, with obesity rates in many large cities approaching or exceeding those in developed countries. The Report on Nutrition and Chronic Disease Status of Chinese Residents (2020) shows that the overweight and obesity rate among children aged 6-17 in China has approached 20%, with 10% of children under 6 years old. The imbalance between energy intake and expenditure is the direct cause of individual overweight and obesity. The 2021 "Healthy Children Action Plan (2021-2025)" explicitly requires the implementation of early screening, early diagnosis, and early treatment prevention and control strategies for risk factors such as obesity that seriously endanger children's health, reducing disease burden, promoting children's health, emphasizing the principle of prevention first and combining prevention and treatment. Given the current status of children's nutrition and health in China, it is an urgent need to establish a standardized and regulated monitoring and management system for obesity and overweight in preschool children, as well as service standards, for the development of children's health. This project aims to establish a complete prevention, improvement, and intervention promotion plan for obesity and overweight in preschool children, as well as a comprehensive monitoring and management system that combines medicine, education, home, and community. It will strengthen children's nutrition feeding and exercise guidance, reduce sedentary time, promote food and movement balance, and prevent and reduce childhood overweight and obesity. Provide children with comprehensive, full process, and warm children's healthcare clothing, and provide small-scale policy research references for the implementation of support systems for children's nutrition improvement projects.

DETAILED DESCRIPTION:
1. Procedures. Step 1: Epidemiological survey: Conduct a health survey on preschool children in selected kindergartens to understand the prevalence and risk factors of overweight and obese children; Phase 2: Recruit overweight and obese children from kindergartens with a population of over 200 in Chongqing, and randomly divide them into an intervention group and a blank control group. Dietary and exercise management, combined with reward and support mechanism monitoring, were implemented for the intervention group, while the blank control group did not receive the aforementioned interventions. Measure the height, weight, BMI, questionnaire survey, blood indicators, etc. of the children before and after the intervention, and use them as evaluation indicators.
2. The sample size for comparing the means of the two groups is N=(Z α/2+Z β) 2 σ 2 (Q1-1+Q2-1)/δ 2. If the difference in BMI decrease between the two groups after intervention is 0.58, and if σ=1.2 and α is taken as 0.05 on both sides, the test power is 0.8, Q1=Q2=0.5，σ=1.2，δ=0.58，Z0.05/2=1.96，Zβ=0.842， Calculate N=(1.96+0.842) 2 * 1.22 * (0.5-1+0.5-1)/0.582 ≈ 69, taking into account the situation of loss to follow-up and refusal to follow up at 20%. The final required two groups of research subjects are 87, and a total of at least 174 research subjects will be included.

4. Statistical analysis. SPSS 26.0 software was used for statistical analysis, and descriptive statistics were performed on general demographic data. Count data was expressed as n (%), and inter group comparisons of rates were performed using a 2-test. Continuous variables that followed a normal distribution were described as mean ± standard deviation (x ± s), and inter group comparisons were performed using t-test. All tests were two-sided, and the test level α was set to 0.05. Multivariate logistic regression analysis of the correlation between nutritional status and risk factors. Using rank sum test to compare the differences in various indicators before and after intervention in obese and overweight children.

5.Ethical matters and data protection. The patients participated in the study will sign the informed consent (obtained from the guardian). And this study was approved by the local ethics committee. Patient's name will be abbreviated and the research data will be assigned a code then to provide to the researcher. The authorization from parents on the patient's health information remains valid until the study is completed. After that, researchers will delete private information from the study record.

ELIGIBILITY:
Inclusion Criteria:

overweight or obese Children Currently, there are no projects related to overweight and obesity management (such as weight loss management, etc.) Parents and children are willing to accept dietary and exercise management for a period of 4 months Willing to measure height, weight, BMI, blood pressure, body composition, questionnaire survey (exercise, diet, etc.) and other items before intervention and 1 month, 2 months, 3 months, and 4 months after intervention (a total of 5 times) Willing to undergo blood tests before and 4 months after intervention (2 times in total); The questionnaire information is filled in accurately and meets the questionnaire quality control standards

Exclusion Criteria:

Recruiter exclusion criteria:

Preschool children with underlying diseases (such as congenital heart disease, liver and kidney disease, thyroid disease, malignant tumors, etc.) or uncontrolled underlying diseases

Questionnaire exclusion criteria:

Incorrect information filling in the questionnaire, which does not meet the questionnaire quality control standards

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 174 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
BMI | 3-4 months
  Changes in BMI between the experimental group and intervention group at the beginning and end of the project

SECONDARY OUTCOMES:
Body composition--Fat (%) | 3-4 months
  Changes in Body composition including Fat (%) between the experimental group and intervention group at the beginning and end of the project.
Body composition--Body fat index (BFMI) | 3-4 months
  Changes in Body composition including Body fat index (BFMI) between the experimental group and intervention group at the beginning and end of the project.
Body composition--Fat-free mass index (FFMI) | 3-4 months
  Changes in Body composition including Fat-free mass index (FFMI) between the experimental group and intervention group at the beginning and end of the project.

OTHER OUTCOMES:
questionnaire investigation | 3-4 months
  Changes in questionnaire investigation（involving diet, exercise, and obesity awareness） between the experimental group and intervention group at the beginning and end of the project
Blood indicators--ALT | 3-4 months
  Changes in blood indicators including glutamic-pyruvic transaminase (ALT) between the experimental group and intervention group at the beginning and end of the of the project.
Blood indicators--AST | 3-4 months
  Changes in blood indicators including glutamic-oxaloacetic transaminase(AST) between the experimental group and intervention group at the beginning and end of the of the project.
Blood indicators--creatinine | 3-4 months
  Changes in blood indicators including creatinine between the experimental group and intervention group at the beginning and end of the of the project.
Blood indicators--uric acid | 3-4 months
  Changes in blood indicators including uric acid between the experimental group and intervention group at the beginning and end of the of the project.
Blood indicators--urea | 3-4 months
  Changes in blood indicators including urea between the experimental group and intervention group at the beginning and end of the of the project.
Blood indicators--blood sugar | 3-4 months
  Changes in blood indicators including blood sugar between the experimental group and intervention group at the beginning and end of the of the project.
Blood indicators--triglyceride | 3-4 months
  Changes in blood indicators including triglyceride between the experimental group and intervention group at the beginning and end of the of the project.
Blood indicators--cholesterol | 3-4 months
  Changes in blood indicators including cholesterol between the experimental group and intervention group at the beginning and end of the of the project.
Blood indicators--high-density | 3-4 months
  Changes in blood indicators including high-density lipoprotein between the experimental group and intervention group at the beginning and end of the of the project.
Blood indicators--low density lipoprotein | 3-4 months
  Changes in blood indicators including low density lipoprotein between the experimental group and intervention group at the beginning and end of the of the project.
Blood indicators--VD | 3-4 months
  Changes in blood indicators including VD between the experimental group and intervention group at the beginning and end of the of the project.
Blood indicators--VA | 3-4 months
  cators including VA between the experimental group and intervention group
Blood indicators--ferritin | 3-4 months
  cators including ferritin between the experimental group and intervention group

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Growth,Development and Mental Health of Children and Adolescents Center, Chongqing, Chongqing Municipality
  - Children's Hospital of Chongqing Medical University, Chongqing

IPD SHARING:
Plan to Share IPD: No
Data is confidential during the study.

REFERENCES:
- [Background] Dong YH, Chen L, Liu JY, Ma T, Zhang Y, Chen MM, Zhong PL, Shi D, Hu PJ, Li J, Dong B, Song Y, Ma J. [Epidemiology and prediction of overweight and obesity among children and adolescents aged 7-18 years in China from 1985 to 2019]. Zhonghua Yu Fang Yi Xue Za Zhi. 2023 Feb 28;57:11-19. doi: 10.3760/cma.j.cn112150-20220906-00881. Online ahead of print. Chinese. PMID 36854438
- [Background] Lister NB, Baur LA, Felix JF, Hill AJ, Marcus C, Reinehr T, Summerbell C, Wabitsch M. Child and adolescent obesity. Nat Rev Dis Primers. 2023 May 18;9(1):24. doi: 10.1038/s41572-023-00435-4. PMID 37202378
- [Result] Hughes AR, Sherriff A, Ness AR, Reilly JJ. Timing of adiposity rebound and adiposity in adolescence. Pediatrics. 2014 Nov;134(5):e1354-61. doi: 10.1542/peds.2014-1908. Epub 2014 Oct 13. PMID 25311600
- [Result] Brown T, Moore TH, Hooper L, Gao Y, Zayegh A, Ijaz S, Elwenspoek M, Foxen SC, Magee L, O'Malley C, Waters E, Summerbell CD. Interventions for preventing obesity in children. Cochrane Database Syst Rev. 2019 Jul 23;7(7):CD001871. doi: 10.1002/14651858.CD001871.pub4. PMID 31332776